CLINICAL TRIAL: NCT04212871
Title: The Effect of Mukbang on the Desire to Eat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1901008509
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Mukbang
Keywords: mukbang; desire to eat

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- watch mukbang (Experimental): In the online study, participants were assigned to watch a ramen mukbang, by Yuka Kinoshita (https://youtu.be/ArPaid2Iuck, accessed: 2018-10-12).
  In the in-person study, participants were assigned to watch a hotpot mukbang by Alun (https://youtu.be/QCTOo9UGZD8, accessed: 2018-11-29).
  Interventions: Other: watch food video 1
- watch another food content video (Experimental): In the online study, participants were assigned to watch a donut mukbang, by Yuka Kinoshita (https://youtu.be/ntMT2y0MgHk, accessed: 2018-10-12).
  In the in-person study, participants were assigned to watch a hotpot cooking show by the Cat's kitchen (https://youtu.be/EH5Ei-sMP60, accessed: 2018-11-29).
  Interventions: Other: watch food video 2
- watch a non-food content video (Placebo Comparator): In the online study, participants were assigned to watch a silent documentary introducing the Palace Museum by China Central Television (CCTV) (https://youtu.be/hWnm1BQOTZY, accessed: 2018-10-12).
  In the in-person study, participants were assigned to watch a video introducing Cornell University is used for the non-food content video (https://youtu.be/GuM8vTq0jd4, accessed: 2018-11-29).
  Interventions: Other: watch a non-food content video

INTERVENTIONS:
Other: watch food video 1 — A 2 minutes video, with food content. The first study used a ramen mukbang here, the second study used a hotpot mukbang.
  Arms: watch mukbang
Other: watch food video 2 — A 2 minutes video, with food content (different content from video 1). The first study used a donut mukbang here, the second study used a hotpot cooking show here.
  Arms: watch another food content video
Other: watch a non-food content video — a 2 minutes video without food content. The first study used a documentary introducing the forbidden city, the second study used a documentary introducing Cornell University.
  Arms: watch a non-food content video

SUMMARY:
Mukbang is an online eating broadcast where a host (Asian mukbangs generally feature a young and slim female host) consumes a large amount of food while chatting with audiences. Since some dieters watch mukbang to get satiation and control their appetites, the current study is aimed at testing the effect of mukbang on the desire to eat.

Two randomized and controlled trails are conducted. The first randomized and controlled trail is conducted online using the Amazon Mturk. Participants (n=286) were randomly assigned to watch one of the following 3 videos: ramen mukbang (n=98), donut mukbang (n=97) and a non-food content video (n=91). The other study is a in person study. Participants (n=234) were randomly assigned to watch one of the following 3 videos: hotpot mukbang (n=79), hotpot cooking show (n=76) and a non-food content video (n=79).

The investigators used the self-report survey to test whether the mukbang affects the desire to eat, and participants' satiation and disgust.

ELIGIBILITY:
Inclusion Criteria:

* Female, age at least 18

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
satiation | immediately after the intervention (after watching the video)
  participants evaluate their satiation level on a scale from -3 to 3. -3 means not satisfied at all, 3 means very satsfied.
disgust | immediately after the intervention (after watching the video)
  participants evaluate their disgust level on a scale from -3 to 3. -3 means not disgust at all, 3 means very disgust.
pre-video desire to eat food | before watching the video. Evaluating the desire to eat was the first step in the study. After reporting this pre-video desire to eat, participants then watched the video.
  participants evaluate their desire to eat food on a scale from 0 to 10. 0 means not want to eat food at all, 10 means very want to eat the food.
post-video desire to eat food | immediately after watching the video. After watching the video, participants immediately re-evaluated their desire to eat, which is this post-video desire to eat.
  participants evaluate their desire to eat food on a scale from 0 to 10. 0 means do not want to eat food at all, 10 means very want to eat the food.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided